CLINICAL TRIAL: NCT01438034
Title: Kisspeptin in the Evaluation of Delayed Puberty
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Stephanie B. Seminara, MD, Chief, Reproductive Endocrine Unit; Professor of Medicine, Harvard Medical School; Director, MGH Harvard Center for Reproductive Medicine, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2011P002885
Record Dates: First submitted 2011-08-24; First posted 2011-09-21 (Estimated); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Delayed Puberty; Kallmann Syndrome; Hypogonadotropic Hypogonadism; GnRH Deficiency
Keywords: delayed puberty; Kallmann Syndrome; Hypogonadotropic hypogonadism; GnRH Deficiency; kisspeptin; GnRH
MeSH Terms: conditions — Puberty, Delayed; Kallmann Syndrome; Hypogonadism | interventions — Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Kisspeptin, GnRH (Experimental): Intravenous (IV) administration of kisspeptin 112-121 0.24 nmol/kg and GnRH 75 ng/kg
  Interventions: Drug: kisspeptin 112-121; Drug: GnRH

INTERVENTIONS:
Drug: kisspeptin 112-121 — 0.24 nmol/kg
  Other Names: metastin 45-54
Drug: GnRH — 75 ng/kg

SUMMARY:
The goal of this study is to test whether the hormone kisspeptin has the potential to prospectively diagnose adolescents with self-resolving or permanent delayed puberty. Some children with delayed puberty will eventually enter puberty on their own. However, some children with delayed puberty have a permanent condition and require medical treatment to undergo puberty. Right now, there is no reliable diagnostic tool to tell whether a child's delayed puberty will be self-resolving or permanent. The hormone kisspeptin has the potential to prospectively diagnose adolescents with self-resolving or permanent delayed puberty.

DETAILED DESCRIPTION:
The investigators are seeking boys (ages 13.5-17 years) and girls (ages 12-17) years with a diagnosis of delayed puberty. Study participation involves 2 outpatient visits and two hospital admissions (one 11-hour, overnight admission and one 6-hour day admission) when subjects will receive two investigational drugs, the naturally occurring hormones kisspeptin and gonadotropin-releasing hormone (GnRH). Subjects will then be followed every 6 months until they reach 18 years of age to determine if their pubertal delay was self-resolved or permanent.

ELIGIBILITY:
Inclusion Criteria:

Adolescent Boys

* ages 13.5-17 years
* testicular volume <4 mL OR 4-8 ml with no change in the past 6 months by Prader orchidometer
* first morning (before 9AM) LH <2 mIU/mL and testosterone <50 ng/dL

Adolescent Girls

* ages 12-17 years
* Tanner stage I OR II breast development with no change in the past 6 months
* first morning (before 9AM) LH <2 mIU/mL and estradiol <20 pg/ml

All Subjects:

* bone age less than chronological age
* weight ≥ 28 kg
* body mass index >10th percentile and <+3 SDS for bone age
* blood pressure >5th percentile and <95th percentile for bone age and height
* white blood cell counts, platelet counts, electrolytes, thyroid stimulating hormone (TSH), free thyroxine (T4) within reference range for age
* erythrocyte sedimentation rate <2X the upper limit of the reference range for age
* hemoglobin within reference range for girls of the same chronological age
* blood urea nitrogen (BUN), creatinine, prolactin not elevated
* aspartate aminotransferase (AST) and alanine aminotransferase (ALT) no more than 2X the upper limit of the reference range
* Insulin-like growth factor 1 (IGF-1) within reference range for bone age

Exclusion Criteria:

All Subjects:

* history or presence of underlying condition that could cause delayed puberty (chronic illness, weight loss, abnormal cranial magnetic resonance imaging (MRI))
* history of an allergic drug reaction

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2013-06-08 (Actual); Primary Completion 2019-09-08 (Actual); Study Completion 2021-09-10 (Actual)

PRIMARY OUTCOMES:
Average change in luteinizing hormone (LH) in response to kisspeptin | Within 30 minutes of administration

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie B Seminara, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chan YM, Lippincott MF, Sales Barroso P, Alleyn C, Brodsky J, Granados H, Roberts SA, Sandler C, Srivatsa A, Seminara SB. Using Kisspeptin to Predict Pubertal Outcomes for Youth With Pubertal Delay. J Clin Endocrinol Metab. 2020 Aug 1;105(8):e2717-25. doi: 10.1210/clinem/dgaa162. PMID 32232399
- [Derived] Chan YM, Lippincott MF, Kusa TO, Seminara SB. Divergent responses to kisspeptin in children with delayed puberty. JCI Insight. 2018 Apr 19;3(8):e99109. doi: 10.1172/jci.insight.99109. eCollection 2018 Apr 19. PMID 29669934